CLINICAL TRIAL: NCT04775342
Title: Smartphone Dual Tasking and Posture Control In Healthy Adolescents
Brief Title: Smartphone and Posture Control In Healthy Adolescents
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Esraa Abd Elaziz Anter, assistant lecturer, Cairo University
Other Study IDs: smartphone and adolescents
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Balance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1 group: 1 group will be assessed then will be given smartphone to use and assessed
  Interventions: Device: smartphone

INTERVENTIONS:
Device: smartphone — modern technology
  Other Names: touch screen

SUMMARY:
This is a study to determine if smartphone use affect posture control in adolescents.

DETAILED DESCRIPTION:
It is within subject repeated measure study to determine if touch screen use affect posture control in healthy adolescents.

200 normal adolescents between 14 and 18 years old will be included.

1st they will be assessed for posture control to determine normal values for their ages, then each child will be given smartphone to play a game while the sound is muted for 15 min then their balance will be re-assessed, finally they will use the phone for another 15 min but the children will use headphone piece this time then re-assess balance.

ELIGIBILITY:
Inclusion Criteria:

* Children age from 14 to 18 years old.
* Both genders will be included.
* Normal Body mass index (BMI) for age.
* Children using smartphone for at least 1 year.

Exclusion Criteria:

* Obese children.
* children with vestibular or visual problems.
* Children with neurological disorders.
* Children with congenital deformities or musculoskeletal disorders.
* Children with cognitive impairment.
* Injuries or inflammatory conditions involving the extremities.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Normal Adolescents
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-11-27 (Actual)

PRIMARY OUTCOMES:
center of pressure | 6 months
  a metric for measuring changes in posture control

CONTACTS AND LOCATIONS:
Overall Officials: Amira M Eltohamy, Study Chair — professor at Cairo university
Locations (1):
- Esraa Abd Elaziz Anter Abd Elaziz, Cairo, Egypt